CLINICAL TRIAL: NCT03028818
Title: An Observational Study of the Epidemiology of Fever Due to Infection in Critically Ill Children Following an Unplanned Admission to a Paediatric Intensive Care Unit
Brief Title: Fever Observational Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Intensive Care National Audit & Research Centre (Other)
Collaborators: Institute of Child Health (Other); Paediatric Intensive Care Audit Network (PICANet) (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 209929
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To inform the feasibility of conducting a study to test different temperature thresholds at which clinicians deliver interventions to reduce fever (i.e. antipyretic interventions) in critically ill children with fever due to infection.

DETAILED DESCRIPTION:
Fever (high temperature) is a normal bodily response to an infection, which has shown to have a beneficial effect in humans with chickenpox, malaria and rhinovirus infections. In children it has been recommended by the National Institute for Health and Care Excellence not to cool down the child using drugs or physical methods such as a cooling mat, with the sole aim to reducing the child's temperature. However, this recommendation is not aimed at the management of critically ill children, to which there is uncertainty around use of cooling interventions when considering the advantages of a fever in defending the body against viruses and bacteria during critical illness, and weighing that up with the possible negative physiological consequences of a high fever e.g. increased metabolic rate.

Observational studies show that the treatment of fever in critically ill children is inconsistent. There is a lack of robust data to guide antipyretic intervention, with clinicians usually starting fever management at around 37.5°C. Evidence is emerging that fever may be beneficial in critically ill adults. Due to the physiological differences between adults and children there is an important need to evaluate whether a different approach to fever management in critically ill children may also be beneficial.

Prior to conducting a large, expensive, randomised clinical trial (RCT) to evaluate whether a higher temperature threshold in starting treatments to cool down the child would be beneficial, we are conducting three studies to know if it is possible for us to test key outcome measures as a result of testing different temperatures thresholds for antipyretic management.

The Fever Observational Study is one of these studies, with the aim of identifying: the potential population that would be eligible for the proposed definitive trial, current temperature threshold(s) for fever management, and to describe the characteristics of outcome measures with the intention of deciding on a main measure to see which treatment method was more successful.

ELIGIBILITY:
Inclusion Criteria:

unplanned PICU admission referral requiring PICU admission to a participating unit

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All unplanned admissions to a PICU
Sampling Method: Non-Probability Sample
Enrollment: 3960 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
To determine the number of patients who meet the eligibility criteria for a proposed definitive trial. | Baseline
Temperature thresholds currently employed in at least 20 paediatric intensive care units (PICU) in the UK | First 5 calender days
Length of ventilation - mean (standard deviation) | Through study completion, an average of 2 days
Length of PICU stay - mean (standard deviation) | Through study completion, an average of 2 days
PICU mortality - number (percentage) | Through study completion, an average of 2 days
Hospital mortality - number (percentage) | Through study completion, an average of 2 days
Days of organ specific support - mean (standard deviation) | Through study completion, an average of 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Peters, MBChB, PhD, Principal Investigator — Institute of Child Health
Locations (1):
- Intensive Care National Audit and Research Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deja E, Peters MJ, Khan I, Mouncey PR, Agbeko R, Fenn B, Watkins J, Ramnarayan P, Tibby SM, Thorburn K, Tume LN, Rowan KM, Woolfall K. Establishing and augmenting views on the acceptability of a paediatric critical care randomised controlled trial (the FEVER trial): a mixed methods study. BMJ Open. 2021 Mar 10;11(3):e041952. doi: 10.1136/bmjopen-2020-041952. PMID 33692177
- [Derived] Peters MJ, Khan I, Woolfall K, Deja E, Mouncey PR, Wulff J, Mason A, Agbeko R, Draper ES, Fenn B, Gould DW, Koelewyn A, Klein N, Mackerness C, Martin S, O'Neill L, Ramnarayan P, Tibby S, Tume L, Watkins J, Thorburn K, Wellman P, Harrison DA, Rowan KM. Different temperature thresholds for antipyretic intervention in critically ill children with fever due to infection: the FEVER feasibility RCT. Health Technol Assess. 2019 Feb;23(5):1-148. doi: 10.3310/hta23050. PMID 30793698